CLINICAL TRIAL: NCT06089070
Title: Feasibility of the FreeStyle Libre Continuous Glucose Monitoring System in Youth With Type 2 Diabetes (FREE CGM)
Brief Title: Continuous Glucose Monitoring System Feasibility in Youth With T2D
Acronym: FREE CGM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-38272
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes
Keywords: freestyle libre; continuous glucose monitor; type 2 diabetes; T2D; pediatric
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Feasibility study of the FreeStyle Libre Continuous Glucose Monitoring System in Youth with Type 2 Diabetes
Masking Description: N/A both study team and participants will know the randomization assignment as to which group they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control (No Intervention): Participants will not have access to view the data from the CGM sensor during the screening period, nor during the main part of the study.
- Intervention (Experimental): Participants will wear the CGM sensor and have access to the data during the main part of the study.
  Interventions: Device: FreeStyle Libre Continuous Glucose Monitor System

INTERVENTIONS:
Device: FreeStyle Libre Continuous Glucose Monitor System — Continuous Glucose Monitor System for people with Type 2 Diabetes
  Arms: Intervention

SUMMARY:
The primary scientific question of this proposal is to investigate whether youth with T2D will wear and interact with a continuous glucose monitor (CGM) system and whether this will influence behavior and management decisions. There will be 30 participants enrolled in the study. 20 in the treatment arm and 10 in the control. The length of study participation will be 6 months for each participant.

DETAILED DESCRIPTION:
At the beginning of the study, participants will be asked to complete surveys where demographic, clinical and behavioral data will be collected. We will ask participants to wear a glucose sensor that is "blinded" for 14-days so that we can gather baseline data about blood sugar levels.

Participants must wear the CGM sensor for at least 10 days out of the 14 days of the blinding period to move on to the next part of the study. After wearing the blinded sensor, the study team will place participants in one of two groups:

One group (intervention group) will be shown how to use the sensors along with the FreeStyle Libre App, and the other group (control group) will continue with their standard diabetes care without using the CGM system. Participants will be "randomized" into one of the study groups described below. Participants will have a 2 in 3 chance of being placed in the group who receives the glucose sensor and will have access to the data.

Group 1 participants will receive the FreeStyle Libre 3 sensor and have access to the data on their smartphone during the study.

Group 2 participants will be asked to continue standard blood glucose monitoring with a glucometer. Participants will be asked to perform 2 checks a day, fasting and 2 hours post dinner as is standard practice.

If randomized to group 1, participants will receive the FreeStyle Libre 3 system with education from the study coordinator on how to insert sensors and view data on the connected mobile app.

Standardized study education materials with suggestions on how to react to the data such as avoidance of sugary beverages or increased physical activity will also be provided.

Participants will be asked to wear the sensor for the rest of the 6-month participation in the study.

If randomized to group 2, participants will be asked to continue standard blood glucose monitoring with a glucometer. Participants will also receive standardized study education materials about reacting to glucose values. Participants will be asked to perform 2 glucose checks a day, fasting and 2 hours after a meal as is standard practice.

As a part of usual care, participants will come to clinic 3 months after starting the study to meet with their usual diabetes provider and a diabetes educator. We will also have a phone check-in visit with participants at 1 month, 2 months, 4 months, and 5 months after starting the study.

For month 3 and month 6 of the study, participants will already be in clinic to see their regular diabetes provider and we can combine their clinic and research visit. At the end of the study, participants will be invited to come to an optional online focus group to talk about the technology that you used with the study researchers.

Participants will be able to share the things that they liked or did not like about the technology. The researchers will speak with approximately 5-7 participants at a time in a group. The conversation will be recorded via a secure videoconference so that the researchers can remember everything that was said. The audio files will be stored in secure locations and participants' full names will not be used in the sessions.

Additional notes:

* If participants do not have the appropriate device to download the app, a reader will be provided by the study team.
* Diagnoses, medication history, medical history, and lab results will be collected from the medical record for research purposes.
* A Random number generator will be used for randomization.
* The study coordinators and/or the investigators will distribute the participant surveys.
* The study coordinators and the investigators will conduct the focus groups.
* There are no in patient procedures.
* For younger participants who may not be able to complete surveys by themselves, parents or guardians may assist younger participants to complete the surveys.

Parents will be requested to complete the parent reports.

ELIGIBILITY:
Inclusion Criteria:

1. Age 8- 20 years at the time of consent.
2. Clinical diagnosis of type 2 diabetes.
3. Duration of type 2 diabetes at least 4 weeks.
4. HbA1C ≥ 6.5% .
5. Stable medication regimen (No medication changes and no change in basal insulin dose by more than 20% in the 2 weeks prior to enrollment).
6. No use of CGM 90 days before screening visit.
7. English or Spanish speakers.
8. Willing to abide by recommendations and study procedures.
9. Willing and able to sign the Informed Consent Form (ICF) and/or has a parent or guardian willing and able to sign the ICF.
10. Participant and parent(s)/guardian(s) willingness to participate in all training sessions as directed by study staff. Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

1. Pancreatic autoantibody positivity (GAD-65, insulin, IA-2, ICA 512, Zn-T8).
2. Plan for undergoing bariatric surgery during the study period.
3. Known history of significant mental illness or developmental delay impacting the ability to complete study activities independently.
4. Known history of adrenal insufficiency, or ongoing renal or hepatic disease.
5. Pregnancy or lactation.
6. Currently undergoing cancer treatment or systemic treatment with steroids.
7. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Ability to use CGM | Measured at 6 months
  Use of CGM measured by number of hours participants in the intervention arm wear the CGM device and view data on the mobile application.
Acceptability of CGM use measured with Acceptability of Intervention Measure (AIM) | Measured at 6 months
  The perception that CGM use is agreeable or satisfactory measured with the 4-item Acceptability of Intervention Measure (AIM). Greater the score, higher the acceptability
Appropriateness of CGM use measured with Intervention Appropriateness Measure | Measured at 6 months
  The perceived fit of the CGM to improve diabetes related metrics measured with the 4-item Intervention Appropriateness Measure (IAM). Greater the score, higher the appropriateness of CGM use
Feasibility of CGM use measured with Feasibility of Intervention Measure. | Measured at 6 months
  The extent to which a CGM study can be successfully carried out measured with 4-item Feasibility of Intervention Measure (FIM). The higher the score, the greater the feasibility of CGM use

SECONDARY OUTCOMES:
Glycemic change | Baseline (0) to 6 months
  Change in HbA1C at 6 months adjusted for the baseline value youth with T2D.
Time in target glucose range | Baseline (0) to 6 months
  Time spent in target glucose range of 70 to 180 mg/dL
Time above high glucose range | Baseline (0) to 6 months
  percent of readings and time >250 mg/dL
Time above glucose range | Baseline (0) to 6 months
  percent of readings and time 181-250 mg/dL
Time below glucose range | Baseline (0) to 6 months
  percent of readings and time 54-69 mg/dL
Time below low glucose range | Baseline (0) to 6 months
  percent of readings and time <54 mg/dl
Glucose management indicator | Baseline (0) to 6 months
  CGM metric that indicates average blood glucose
Co-efficient of variation of glucose | Baseline (0) to 6 months
  CGM metric that measures variability in CGM values
Change in BMI | Baseline (0) to 6 months
  Change in BMI SDS over the course of the study
Frequency of taking diabetes medications | Baseline (0) to 6 months
  Self-reported medication adherence in the past week before visit
Starting or stopping medications | Baseline (0) to 6 months
  Percentage of subjects with addition or removal of diabetes medications
Titration of insulin dosing by provider | Baseline (0) to 6 months
  Percentage of subjects who receive insulin dose titration
Dietary measures | Baseline (0) to 6 months
  Change in score on SEARCH for Diabetes in Youth food frequency questionnaire. This is a 85 question survey ( Mayer-Davis EJ, Nichols M, Liese AD et al. (2006) Dietary intake among youth with diabetes: the SEARCH for Diabetes in Youth Study. J Am Diet Assoc.2006)
Physical activity measures | Baseline (0) to 6 months
  Number of minutes of physical activity in the past week before visit. The greater the value the better the score.
Quality of Life score on survey | Baseline (0) to 6 months
  Pediatric Quality of Life Inventory Diabetes Module score. 33 item score. The greater the value the better the score.
Problem Areas in Diabetes | Baseline (0) to 6 months
  Problem Areas In Diabetes (PAID) Scale. 20 question survey. Higher the score, the worse the outcome

CONTACTS AND LOCATIONS:
Overall Officials: Shylaja Srinivasan, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco (UCSF), San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wagenknecht LE, Lawrence JM, Isom S, Jensen ET, Dabelea D, Liese AD, Dolan LM, Shah AS, Bellatorre A, Sauder K, Marcovina S, Reynolds K, Pihoker C, Imperatore G, Divers J; SEARCH for Diabetes in Youth study. Trends in incidence of youth-onset type 1 and type 2 diabetes in the USA, 2002-18: results from the population-based SEARCH for Diabetes in Youth study. Lancet Diabetes Endocrinol. 2023 Apr;11(4):242-250. doi: 10.1016/S2213-8587(23)00025-6. Epub 2023 Feb 28. PMID 36868256
- [Result] TODAY Study Group; Bjornstad P, Drews KL, Caprio S, Gubitosi-Klug R, Nathan DM, Tesfaldet B, Tryggestad J, White NH, Zeitler P. Long-Term Complications in Youth-Onset Type 2 Diabetes. N Engl J Med. 2021 Jul 29;385(5):416-426. doi: 10.1056/NEJMoa2100165. PMID 34320286
- [Result] TODAY Study Group; Zeitler P, Hirst K, Pyle L, Linder B, Copeland K, Arslanian S, Cuttler L, Nathan DM, Tollefsen S, Wilfley D, Kaufman F. A clinical trial to maintain glycemic control in youth with type 2 diabetes. N Engl J Med. 2012 Jun 14;366(24):2247-56. doi: 10.1056/NEJMoa1109333. Epub 2012 Apr 29. PMID 22540912
- [Result] U.K. prospective diabetes study 16. Overview of 6 years' therapy of type II diabetes: a progressive disease. U.K. Prospective Diabetes Study Group. Diabetes. 1995 Nov;44(11):1249-58. PMID 7589820